CLINICAL TRIAL: NCT04418102
Title: The InterSat Study: Interesterified Fats: Health Effects of Commercially Relevant Palmitic Versus Stearic Acid Rich Interesterified Fats
Brief Title: The InterSat Study
Acronym: InterSat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HR-19/20-14655
Record Dates: First submitted 2020-02-19; First posted 2020-06-05 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Cardiometabolic Health
Keywords: Interesterified fat; Cardiometabolic health; Palmitic acid; Stearic acid; Vascular function; Postprandial lipaemia

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with 2x6 week interventions separated by a 3 week washout.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palmitic acid rich interesterified fat (Experimental): Snacks (muffins) and spread containing palmitic acid rich interesterified fat to replace habitual snacks and spreads, and provide 10% of total daily energy intake with the interesterified fat.
  Interventions: Dietary Supplement: Palmitic acid rich interesterified fat
- Stearic acid rich interesterified fat (Active Comparator): Snacks (muffins) and spread containing stearic acid rich interesterified fat to replace habitual snacks and spreads, and provide 10% of total daily energy intake with the interesterified fat.
  Interventions: Dietary Supplement: Stearic acid rich interesterified fat

INTERVENTIONS:
Dietary Supplement: Palmitic acid rich interesterified fat — Muffins and spread containing the palmitic acid rich IE fat will be consumed daily for a 6-week dietary intervention period
  Arms: Palmitic acid rich interesterified fat
Dietary Supplement: Stearic acid rich interesterified fat — Muffins and spread containing the palmitic acid rich IE fat will be consumed daily for a 6-week dietary intervention period.
  Arms: Stearic acid rich interesterified fat

SUMMARY:
In response to the removal of trans fats from our foods, the food industry now uses interesterified (IE) fats. Randomly interesterified (IE) fats rich in palmitic (Europe) and stearic (North America) acids are the most commonly used IE fats by the food industry. Despite their widespread use, there has been no published research on the acute and chronic cardio-metabolic health effects of the most commonly consumed palmitic and stearic acid rich IE fats. The aim of InterSat is to investigate the postprandial and chronic effects of a diet rich in IE fats on cardiometabolic health.

DETAILED DESCRIPTION:
Choice of design: A randomised crossover study with two arms, each arm consisting of a 6-week dietary intervention, separated by a 3-week (minimum) washout period.

Study population: Healthy adult snackers aged 35-65 years. 48 participants in total, 24 at each centre (see Locations).

Locations:

Metabolic Research Unit, Franklin-Wilkins Building, Waterloo Campus, King College London.

Metabolic Research Unit Maastricht, Academic Hospital Maastricht, Maastricht University.

Screening Assessment: Prospective participants will be selected based on the defined inclusion and exclusion criteria by the study management team. Recruitment will be done over the phone and via the Internet and emails and prospective participants will be booked in for their initial appointment to acquire baseline measurements.

Study duration: A 2-week run-in period, two 6-week dietary interventions, and a 3-week (minimum) washout period.

Dietary intervention: The InterSat intervention aims to provide 10% of total daily energy intake in the form of IE fat. These will be consumed in the form of muffins and spreads, designed to replace typically consumed snacks and spreads throughout the day. Energy requirements will be calculated using the Henry equation and physical activity levels (PAL).

At the baseline visit, participants will have and anthropometric measures and fasted blood samples taken, and will be assessed for endothelial function via flow mediated dilation (FMD), after which they will be provided with enough muffins and spread for a 2-week period, as well a study booklet (containing instructions and a diary to log muffin and spread consumption). They will receive guidance on how to incorporate the muffins and spread into their diet. Food collection dates will be set, and participants are then free to leave. At the second visit (first snack collection visit), no physical measures are taken, but the empty tubs and muffin cases are collected, and the study booklet is checked by a researcher to ensure the participant is compliant to the intervention. Any issues should be discussed, and guidance given to increase compliance if necessary. Another snack collection visit is booked. At the end of the 6-week intervention, participants will undergo physical and blood sampling as well as FMD, as with the baseline testing day. After a 3-week (minimum) washout period, the same procedures occur for the other arm of the trial.

Anthropometry: Weight, height, waist and hip circumference, blood pressure, body fat will be taken using standard procedures, in duplicates by a trained researcher at all face to face appointments.

Habitual food intake: Participants will complete the EPIC (European prospective investigation of cancer) food frequency questionnaire at the screening visit. They will also complete three 4-day diet diaries (one at the run-in period and one in each of the dietary intervention periods).

Blood samples: Fasting blood samples will be collected from a superficial antecubital vein via venepuncture before and after each dietary intervention. Postprandial blood samples will be taken via cannulation in a subgroup (see Subgroup below) for an 8-hour postprandial test day.

Participants will be asked to record and monitor the following information:

Amount of muffins and spread consumed (study booklet). Habitual intake (4-day diet diaries).

Subgroup: A subset (n = 24) of participants will undergo a postprandial test day at the baseline and 6-week points of each intervention arm. After baseline samples (anthropometrics, blood samples, FMD) are taken, participants will consume a breakfast containing a large bolus of the IE fat they are assigned to. Blood samples will be taken over an 8-hour testing period and FMD will be taken 2 more times. Liver fat will be assessed via MRI imaging (Maastricht only).

ELIGIBILITY:
Inclusion Criteria:

* Healthy (free of diagnosed diseases listed in exclusion criteria).
* Able to give informed consent.
* Able to give informed consent.
* Accessible veins on arms as determined by examination at screening

Exclusion Criteria:

* Having a medical condition or history which might impact study measurements, to be judged by the study physician (e.g. myocardial infarction, angina, thrombosis, stroke, cancer, liver or bowel disease or diabetes)
* Use of plant-sterol/stanol-enriched foods or supplements in the three months prior to the screening and/or during the study
* Body mass index < 20 kg/m2 or > 35 kg/m2
* Plasma cholesterol ≥7.5 mmol/L
* Plasma triacylglycerol > 3 mmol/L
* Plasma glucose > 7 mmol/L
* Full blood count (FBC), liver function out of healthy range
* Blood pressure ≥140/90 mmHg
* Current use of antihypertensive or lipid lowering medications
* Use of over-the-counter and prescribed medication, which may interfere with study measurements (to be judged by the principal investigator)
* Alcohol intake exceeding a moderate intake (> 21 units per week)
* Current cigarette smoker (or quit within last 6 months)
* ≥ 20% 10-year risk of cardiovascular disease (CVD) as calculated using a risk calculator
* Active blood donor or plans to donate blood within 6 months of study completion
* Use of oral antibiotics (with the exception of topical antibiotics) in 40 days or less prior to the start of the study
* Reported weight loss or gain of 3 kg or more during a period of 2 months prior to screening
* Reported dietary habits: medically prescribed diet, allergy/intolerance to test products that will be provided during the study
* Reported participation in another nutritional or biomedical trial 3 months prior to screening
* Reported participation in night shift work 2 weeks prior to screening and/or during the study. Night work is defined as working between midnight and 6.00 am Anyone who has given blood in the last 3 months

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fasting total:HDL cholesterol ratio | 6 weeks
  Total to high-density lipoprotein (Total:HDL) cholesterol ratio

SECONDARY OUTCOMES:
Postprandial lipaemia | Fasting, 60 min, 120 min, 180 min, 240 min, 300 min, 360 min, 420 min, 480 min following consumption of breakfast containing IE fats.
  Plasma triglyceride concentrations
Endothelial function | Fasting, 270 min and 450 min following consumption of breakfast containing IE fats
  Flow mediated dilation
Postprandial glucose homeostasis (Incremental area under the curve (iAUC) 0-240 min and 0-480 min) | Fasting, 30 min, 60 min, 120 min, 180 min, 240 min, 300 min, 360 min, 420 min, 480 min following consumption of breakfast containing IE fats.
  Glucose, Insulin, C-peptide, Non-esterified fatty acids (NEFA)
Fasting Insulin sensitivity | Fasting, 30 min, 60 min, 120 min, 180 min, 240 min, 300 min, 360 min, 420 min, 480 min following consumption of breakfast containing IE fats.
  Revised Quantitative Insulin Sensitivity Check Index (RQUICKI)
Change from baseline in liver fat (Maastricht only) | 6 weeks
  MRI (magnetic resonance imaging)
Change from baseline in fasting total cholesterol | 6 weeks
  Fasting plasma total cholesterol concentrations
Change from baseline in fasting LDL cholesterol | 6 weeks
  Fasting plasma low density lipoprotein cholesterol (LDL-C) concentrations
Change from baseline in fasting Lp(a) | 6 weeks
  Fasting plasma lipoprotein a (Lp(a))
Change from baseline in fasting apoA1 | 6 weeks
  Fasting plasma apolipoprotein A1 (apoA1),
Change from baseline in fasting apoB | 6 weeks
  Fasting plasma apolipoprotein B (apo B)
Change from baseline in plasma total fatty acid composition | 6 weeks
  Fasting plasma total fatty acid composition
Change from baseline in fasting glucose | 6 weeks
  Fasting plasma glucose concentrations
Change from baseline in fasting insulin | 6 weeks
  Fasting plasma insulin concentrations

CONTACTS AND LOCATIONS:
Locations (2):
- Maastricht University, Maastricht, Netherlands
- Department of Nutritional Sciences, King's College London. Franklin-Wilkins Buiding. Waterloo Campus, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall WL, Wood E, Joris PJ, Smith HA, Creedon A, Maher T, Bruce JH, Mensink RP, Berry SE. The effects of consumption of interesterified fats rich in palmitic acid compared with stearic acid on intermediary markers of cardiometabolic disease risk: a randomized controlled trial in healthy adults. Am J Clin Nutr. 2025 Nov;122(5):1361-1373. doi: 10.1016/j.ajcnut.2025.09.025. Epub 2025 Sep 18. PMID 40975239